CLINICAL TRIAL: NCT01974245
Title: Impact of Treatment With Cholecalciferol on Immunological Markers in Patients With Hypovitaminosis D on Dialysis
Brief Title: Supplementation With Cholecalciferol in Dialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Lilian Cuppari, Afilliate Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNPq473838/2011-7
Record Dates: First submitted 2013-10-08; First posted 2013-11-01 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease
Keywords: Cholecalciferol; Kidney diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 100 drops/week for 12 weeks
  Interventions: Drug: Placebo
- Cholecalciferol (Active Comparator): Drug: Cholecalciferol - 100,000 IU/week
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 100,000 IU/week for 12 weeks
  Other Names: Vitamina D3
  Arms: Cholecalciferol
Drug: Placebo — 100 drops/ week for 12 weeks
  Arms: Placebo

SUMMARY:
Hypovitaminosis D is highly prevalent among patients with chronic kidney disease, especially in those undergoing dialysis. The loss of protein to the dialysis solution seems to contribute significantly to the reduced serum levels of vitamin D in these patients. As a result of the disease and the dialysis procedure, there is high prevalence of chronic inflammation and high risk of infections. There is evidence in other populations, that vitamin D has immunomodulatory effects by stimulating the production of cathelicidin, an antimicrobial peptide and suppressing the production of proinflammatory cytokines. Thus, this study aims to investigate the effects of cholecalciferol supplementation on immunological markers in patients in hemodialysis and peritoneal dialysis with hypovitaminosis D . This is a randomized, double-blind, placebo-controlled trial in which patients who have vitamin D deficiency [25 (OH) D <20 ng / mL] will be allocated to the intervention group (cholecalciferol) or control (placebo). Patients will receive supplemented 100,000 IU / week cholecalciferol a period of 12 weeks. Before and after the intervention will be determined 25(OH)D, cathelicidin, interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α) and C-reactive protein serum. In monocytes, we will evaluate cathelicidin, IL-6 and TNF-α, 25(OH)D receptor and α 1-hydroxylase enzyme expression.

ELIGIBILITY:
Inclusion Criteria:

* 25 (OH) < 20 ng/ml
* Peritoneal dialysis or hemodialysis > 3 months

Exclusion Criteria:

* Use of vitamin D or its analogues, corticosteroids and immunosuppressive
* Peritonitis in the previous month at baseline
* Liver, neoplastic, infectious or autoimmune diseases and positive HIV
* Hypercalcemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Cuppari, PhD, Principal Investigator — Federal University of São Paulo; Marion S Meireles, Master, Principal Investigator — Federal University of São Paulo; Maria A Kamimura, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Meireles MS, Kamimura MA, Dalboni MA, Giffoni de Carvalho JT, Aoike DT, Cuppari L. Effect of cholecalciferol on vitamin D-regulatory proteins in monocytes and on inflammatory markers in dialysis patients: A randomized controlled trial. Clin Nutr. 2016 Dec;35(6):1251-1258. doi: 10.1016/j.clnu.2016.04.014. Epub 2016 Apr 26. PMID 27161894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2012 and May 2014 the patients from Dialysis Unit of the Federal University of São Paulo and Oswaldo Ramos Foundation (São Paulo, Brazil) were screened.
Pre-assignment Details: Patients that have in use of any vitamin D compounds, glucocorticoids, immunosuppressors, or with history of liver failure, intestinal malabsorption, malignance, autoimmune disease, active infection, positive HIV, peritonitis in the last month or elevated serum ionized calcium (>1.40 mmol/L) were not included in the study.
Groups:
- Placebo: 100 drops placebo solution/week
- Cholecalciferol: Cholecalciferol: 100,000 IU/week
Period: Overall Study
Arm/Group | Placebo | Cholecalciferol
Started | 27 | 28
Completed | 18 | 20
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 100 drops/week
- Total: Total of all reporting groups
Arm/Group | Placebo | Cholecalciferol | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.9) | 55.5 (14.2) | 56.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  Brazil | 18 | 20 | 38
Dialysis therapy [Number; unit: participants]
  Peritoneal dialysis | 6 | 9 | 15
  Hemodialysis | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Interleukin-6 at 12 Weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Cholecalciferol
Number analyzed (Participants) | 18 | 20
pg/mL
  Interleukin-6 baseline | 9.0 (5.2) | 8.1 (6.6)
  Interleukin-6 after intervention | 9.6 (5.6) | 4.6 (4.1)

2. Secondary Outcome: Change From Baseline in C-reactive Protein at 12 Weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change From Baseline in Expression in Monocytes of Vitamin D Receptor, α 1-hydroxylase and 24-hydroxylase Enzymes, and Interleukin-6 at 12 Weeks
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Cholecalciferol
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No